CLINICAL TRIAL: NCT07115810
Title: No Prognostic or Molecular Disparity Between Synchronous and Metachronous Metastases in Differentiated Thyroid Cancer: Insight From Middle Eastern Cohort
Status: Completed | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Khawla S. Al-Kuraya, Dr, King Faisal Specialist Hospital & Research Center
Other Study IDs: RAC#2110031
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Differentiated Thyroid Cancer
Keywords: synchronous metastasis; metachronous metastasis; prognosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic DTC
  Interventions: Other: No additional drugs(control Group)

INTERVENTIONS:
Other: No additional drugs(control Group) — No intervention

SUMMARY:
The goal of this observational study is to compare the clinical outcomes, molecular features, and immune profiles of patients with synchronous and metachronous distant metastases in Saudi cohort with well characterized differentiated thyroid cancer. The main question it aims to answer is whether timing of metastasis is associated with distinct prognostic or biological behavior in differentiated thyroid cancer from a large Middle Eastern cohort

ELIGIBILITY:
Inclusion Criteria:

* Synchronous or metachronous distant metastases

Exclusion Criteria:

* Not DTC
* No distant metastases

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with metastatic differentiated thyroid cancer diagnosed at King Faisal Specialist Hospital & Research Centre in Riyadh, Saudi Arabia
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 1988-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Thyroid cancer-specific survival | 5 years

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to local regulations in Saudi Arabia